CLINICAL TRIAL: NCT03073681
Title: Patient-Reported Satisfaction and Spectacle Independence With the ReSTOR 2.5 Combined With the ReSTOR 3.0 IOL in Cataract Surgery
Brief Title: Satisfaction & Spectacle Independence With ReSTOR 2.5 & ReSTOR 3.0 IOLs
Status: Completed | Type: Observational
Sponsor: MDbackline, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: ALC 2.5/3.0 29576247
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Cataract
Keywords: cataract
MeSH Terms: conditions — Cataract | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Historical controls: This group of historical controls makes up patients who have previously undergone cataract surgery with a 3.0 add ReSTOR lens in each eye. This group has already completed a satisfaction questionnaire identical to what will be posed in the 2.5/3.0 add lens group.
- 2.5 and 3.0 add lenses: This group will have undergone cataract surgery at least 2 months before conducting a questionnaire. Patients enrolled in this group had cataract surgery with a 2.5 add ReSTOR lens in one eye and a 3.0 add lens in the other.
  Interventions: Device: Survey

INTERVENTIONS:
Device: Survey — Patients will complete a survey describing their satisfaction with vision after cataract surgery that was performed at least 2 months prior to study enrollment.
  Groups: 2.5 and 3.0 add lenses

SUMMARY:
Patients implanted with the ReSTOR 2.5 multifocal IOL in the dominant eye and the ReSTOR 3.0 in the non-dominant eye have overall satisfaction and spectacle independence at least comparable to that with bilateral implantation of the 3.0 add lens. Glare and haloes and other unwanted visual side effects with this mixed combination of lenses is better than with bilateral 3.0 lenses.

DETAILED DESCRIPTION:
Patients desire spectacle independence for a range of distances, including distance, intermediate, and near. The ReSTOR 2.5 multifocal lens has been designed to allow better uncorrected intermediate vision and reduce glare and haloes compared to previous, higher-add models. However, their impact on overall patient satisfaction, glare & haloes (incidence and impact), and spectacle independence has not been examined with a patient-reported outcome study. Additionally, in clinical practice, many clinicians find that bilateral implantation of ReSTOR 2.5 yields insufficient near vision for about 30% of patients (1). For this reason, many surgeons prefer to implant the ReSTOR 2.5 in one eye (usually the dominant) and the ReSTOR 3.0 in the other eye.

MDbackline is a multi-center patient-reported research engine that has been in use since 2013 for data collection in several patient-reported outcome studies for major industry sponsors. Studies performed with MDbackline have been presented at major meetings and are in press with peer-reviewed journals. The investigators have previously conducted studies of patient satisfaction and spectacle independence with the higher add (3.0) multifocal lens prior to the approval of the ReSTOR 2.5. These data, which include about 85 patients, will be used as historical references. They showed a high degree of satisfaction and spectacle independence but complaints of glare and haloes in as many as 37% of patients ("a fair amount of glare" or more). (2) Since approval of the ReSTOR 2.5, the investigators have clinically observed far fewer complaints of glare/haloes when the lower-add lens is used in at least one eye.

In this study the investigators propose to evaluate patients with the ReSTOR 2.5 lens in one eye and the ReSTOR 3.0 in the other using substantially the same questionnaire in the previous study described above. The investigators plan to compare results of these new data (2.5/3.0 combination) with the previous study data (3.0/3.0).

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with either a ReSTOR 2.5 or 3.0 multifocal within 24 months of the survey administration.
* Patients with otherwise healthy eyes, not exhibiting any significant ocular morbidity that would be expected to influence outcome measures.

Exclusion Criteria:

* Patients with visually significant co-morbidities (corneal, retina, optic nerve disease) that could affect their satisfaction with surgery
* Patients with surgical complications either during or after surgery (capsule tears, iris trauma, decentered IOL, cystoid macular edema, etc.)
* Patients with previous refractive surgery
* Patients with ≥ grade 1 posterior capsule opacity at their last visit

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with healthy eyes and uncomplicated cataract surgery completed at least 2 months before a questionnaire is conducted.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
Overall satisfaction with surgery | at least 2 months after surgery
  Overall satisfaction with surgery, defined as the percentage of patients who report "top box" (5 out of 5) satisfaction with implantation of a 2.5D add ReSTOR implant in the dominant eye and a 3.0D add ReSTOR implant in the non-dominant eye.

CONTACTS AND LOCATIONS:
Overall Officials: John Hovanesian, MD, Principal Investigator — MDbackline, LLC
Locations (1):
- Harvard Eye Associates, Laguna Hills, California, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD.

REFERENCES:
- [Background] Fraunfelder FW. Corneal toxicity from topical ocular and systemic medications. Cornea. 2006 Dec;25(10):1133-8. doi: 10.1097/01.ico.0000240084.27663.fd. PMID 17172885